CLINICAL TRIAL: NCT00558441
Title: Prospective Data Collection in Clinical Cases Where Coronary Plaque Lipid Characterization by IVMRI Was Performed During Diagnostic or Interventional Catheterization Procedures
Brief Title: Prospective Data Collection of IVMRI Cases
Acronym: MIRACLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TopSpin Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCL-1.2-002
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Plaque Lipid Characterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: IVMRI

INTERVENTIONS:
Device: IVMRI — Intra Vascular Magnetic Resonance Imaging
  Other Names: Cathamaran

SUMMARY:
The study purpose is to prospectively collect data for a set of predefined variables in clinical cases where coronary plaque lipid characterization by IVMRI was performed during diagnostic or interventional procedures in order to gather incremental information beyond angiography and other diagnostic modalities.

ELIGIBILITY:
Inclusion Criteria:

* An adult patient ≥ 18 years old.
* The patient, or legal guardian, has been informed of the nature of the study, agrees to its provisions, and has sign the approved informed consent.
* The patient and the treating physician agree to attend the follow-ups as defined in the study protocol.
* Indication for diagnostic and/or interventional procedure.
* Lesions in a native vessels where IVMRI interrogation may provide additional information beyond angiography and other diagnostic tools.

Exclusion Criteria:

* Culprit lesions within 48 hours following STEMI.
* Tortuous vessels, calcified or thrombotic lesions.
* Significant stenosis of an unprotected left main coronary artery.
* IVMRI interrogation of an unprotected left main coronary artery.
* Patients with pacemaker or cardioverter defibrillator.
* The patient is suffering from transplant mediated coronary artery disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-11; Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
LFI - Lipid Fraction Index | 5 years

SECONDARY OUTCOMES:
correlation between LFI and a set of predefined parameters | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William Wijns, Prof., Principal Investigator — OLV Hospital
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel